CLINICAL TRIAL: NCT03941548
Title: A Randomized Parallel-Group Study to Evaluate the Efficacy and Tolerability of Two Dosing Regimens of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: Efficacy and Tolerability Study of Two Dosing Regimens of CTP-543 in Adults With Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP543.2003
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTP-543 12 mg BID (Experimental): Participants received 1 x 12 milligrams (mg) CTP-543 tablet and 1 x CTP-543 matching placebo tablet, twice daily (BID) for 24 weeks.
  Interventions: Drug: CTP-543; Drug: CTP-543 Matching Placebo
- CTP-543 24 mg QD (Experimental): Participants received 24 mg (2 x 12 mg) CTP-543 tablets, once daily (QD) and after 12 hours, received 2 x CTP-543 matching placebo tablets, QD for 24 weeks.
  Interventions: Drug: CTP-543; Drug: CTP-543 Matching Placebo

INTERVENTIONS:
Drug: CTP-543 — Administered as 12 mg tablets.
Drug: CTP-543 Matching Placebo — Administered as tablets to aid treatment masking.

SUMMARY:
This study will evaluate the efficacy and tolerability of once-daily versus twice-daily dosing of CTP-543, in adult patients with chronic, moderate to severe alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation compatible with alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted.
* At least 50% scalp hair loss, as defined by a Severity of Alopecia Tool (SALT) score ≥50, at Screening and Baseline.

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or untreated actinic keratosis on the scalp.
* Treatment with systemic immunosuppressive medications within 3 months of screening or during the study, or biologics within 6 months of screening or during the study.
* Clinical lab results outside the normal range.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Colorado Center for Dermatology and Skin Surgery, Centennial, Colorado
  - ForCare Clinical Research, Tampa, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
- Canada (7):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - Research Toronto, Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 study centers in Canada and the United States from 24 May 2019 to 10 April 2020.
Pre-assignment Details: 94 participants were screened out of which 66 participants who experienced an episode of hair loss due to alopecia areata were enrolled and randomized to receive CTP-543 12 milligrams (mg) twice daily (BID) or CTP-543 24 mg once daily (QD).
Groups:
- CTP-543 12 mg BID: Participants received 1 x 12 mg CTP-543 tablet and 1 x CTP-543 matching placebo tablet, BID for 24 weeks.
- CTP-543 24 mg QD: Participants received 24 mg (2 x 12 mg) CTP-543 tablets, QD and after 12 hours, received 2 x CTP-543 matching placebo tablets, QD for 24 weeks.
Period: Overall Study
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Started | 34 | 32
Safety Population (Safety population included all participants who received at least one dose of study drug. Participants were summarized according to study drug regimen received.) | 34 | 32
mITT Population (Modified Intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug and had at least 1 post-treatment SALT assessment. Participants were summarized according to study drug regimen to which they were randomized.) | 34 | 32
Completed | 33 | 30
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal of Informed Consent due to an Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug. Participants were summarized according to study drug regimen received.
Groups:
- Total: Total of all reporting groups
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.89) | 40.4 (14.20) | 39.6 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 34 | 29 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 4 | 8
  White | 25 | 23 | 48
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Severity of Alopecia Tool (SALT) Score [Mean (Standard Deviation); unit: score on a scale] — The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss).
  score on a scale | 85.77 (19.473) | 87.76 (17.280) | 86.73 (18.328)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Severity of Alopecia Tool (SALT) Score at Week 24
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Relative change (percent change) to baseline is calculated as: 100 x ([baseline SALT score - follow-up SALT score]/baseline SALT score).
Time Frame: Baseline, Week 24
Population: mITT Population included all randomized participants who received at least one dose of study drug and had at least 1 post-treatment SALT assessment. Participants were summarized according to study drug regimen to which they were randomized.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 34 | 32
percent change | 58.44 (34.747) | 51.96 (37.887)

2. Secondary Outcome: Percentage of Participants Achieving at Least a 90%, 75%, and 50% Reduction in SALT Score From Baseline
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Percentage of participants achieving at least a 50%, 75%, 90% relative reduction in SALT score from baseline at Weeks 4, 8, 12, 16, 20, and 24 are reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 34 | 32
percentage of participants
  90% Reduction: Week 4 | 0.0 | 0.0
  90% Reduction: Week 8 | 0.0 | 0.0
  90% Reduction: Week 12 | 8.8 | 6.3
  90% Reduction: Week 16 | 20.6 | 12.5
  90% Reduction: Week 20 | 32.4 | 21.9
  90% Reduction: Week 24 | 32.4 | 31.3
  75% Reduction: Week 4 | 0.0 | 0.0
  75% Reduction: Week 8 | 0.0 | 0.0
  75% Reduction: Week 12 | 14.7 | 18.8
  75% Reduction: Week 16 | 23.5 | 25.0
  75% Reduction: Week 20 | 35.3 | 31.3
  75% Reduction: Week 24 | 38.2 | 34.4
  50% Reduction: Week 4 | 0.0 | 0.0
  50% Reduction: Week 8 | 8.8 | 0.0
  50% Reduction: Week 12 | 32.4 | 31.3
  50% Reduction: Week 16 | 44.1 | 40.6
  50% Reduction: Week 20 | 52.9 | 43.8
  50% Reduction: Week 24 | 61.8 | 53.1

3. Secondary Outcome: Absolute Change From Baseline in SALT Scores at Weeks 4, 8, 12, 16, 20, and 24
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Absolute change equals the difference in SALT measurements (baseline SALT score - follow-up SALT score).
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 34 | 32
score on a scale
  Change from Baseline at Week 4 | 1.95 (4.247) | 3.02 (5.211)
  Change from Baseline at Week 8 | 11.68 (17.674) | 13.61 (15.795)
  Change from Baseline at Week 12 | 26.07 (28.086) | 25.33 (27.874)
  Change from Baseline at Week 16 | 38.83 (30.699) | 31.32 (28.637)
  Change from Baseline at Week 20 | 45.44 (32.169) | 37.78 (31.021)
  Change from Baseline at Week 24 | 48.63 (31.733) | 42.82 (31.470)

4. Secondary Outcome: Relative Change From Baseline in SALT Scores at Weeks 4, 8, 12, 16 and 20
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16 and 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 34 | 32
percent change
  Change from Baseline at Week 4 | 3.12 (7.474) | 3.95 (7.126)
  Change from Baseline at Week 8 | 14.57 (19.800) | 17.24 (19.034)
  Change from Baseline at Week 12 | 32.10 (30.960) | 31.90 (33.820)
  Change from Baseline at Week 16 | 47.20 (34.663) | 39.08 (35.750)
  Change from Baseline at Week 20 | 54.58 (35.582) | 46.24 (37.891)

5. Secondary Outcome: Percentage of Participants With Change in Satisfaction of Hair Coverage From Baseline
Description: Participant satisfaction question was used to assess overall satisfaction with hair coverage, with responses ranging from 1 to 5, as follows: 1 (very dissatisfied), 2 (dissatisfied), 3 (somewhat satisfied), 4 (mostly satisfied), 5 (very satisfied). Higher scores indicate better satisfaction with hair coverage. The percentage of participants with change from Baseline to Weeks 8, 12 and 24 satisfaction level was reported as categories: satisfied to satisfied; satisfied to dissatisfied; dissatisfied to satisfied and dissatisfied to dissatisfied. Data is reported only for participants with change from Baseline in satisfaction level.
Time Frame: Baseline, Weeks 8, 12 and 24
Population: mITT Population included all randomized participants who received at least one dose of study drug and had at least 1 post-treatment SALT assessment. Participants were summarized according to study drug regimen to which they were randomized, with data available for analysis. Number analyzed indicates the number of participants with available data for analysis at the specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 32 | 31
percentage of participants
  Week 8: Satisfied to Satisfied: number analyzed (Participants) | 28 | 29
  Week 8: Satisfied to Satisfied | 3.6 | 0
  Week 8: Satisfied to Dissatisfied: number analyzed (Participants) | 28 | 29
  Week 8: Satisfied to Dissatisfied | 0 | 0
  Week 8: Dissatisfied to Satisfied: number analyzed (Participants) | 28 | 29
  Week 8: Dissatisfied to Satisfied | 39.3 | 44.8
  Week 8: Dissatisfied to Dissatisfied: number analyzed (Participants) | 28 | 29
  Week 8: Dissatisfied to Dissatisfied | 57.1 | 55.2
  Week 12: Satisfied to Satisfied: number analyzed (Participants) | 31 | 31
  Week 12: Satisfied to Satisfied | 6.5 | 0
  Week 12: Satisfied to Dissatisfied: number analyzed (Participants) | 31 | 31
  Week 12: Satisfied to Dissatisfied | 0 | 0
  Week 12: Dissatisfied to Satisfied: number analyzed (Participants) | 31 | 31
  Week 12: Dissatisfied to Satisfied | 35.5 | 67.7
  Week 12: Dissatisfied to Dissatisfied: number analyzed (Participants) | 31 | 31
  Week 12: Dissatisfied to Dissatisfied | 58.1 | 32.3
  Week 24: Satisfied to Satisfied: number analyzed (Participants) | 32 | 30
  Week 24: Satisfied to Satisfied | 6.3 | 0
  Week 24: Satisfied to Dissatisfied: number analyzed (Participants) | 32 | 30
  Week 24: Satisfied to Dissatisfied | 0 | 0
  Week 24: Dissatisfied to Satisfied: number analyzed (Participants) | 32 | 30
  Week 24: Dissatisfied to Satisfied | 68.8 | 70.0
  Week 24: Dissatisfied to Dissatisfied: number analyzed (Participants) | 32 | 30
  Week 24: Dissatisfied to Dissatisfied | 25.0 | 30.0

6. Other Pre Specified Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event is any untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the patient's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an adverse event.
Time Frame: From first dose up to 28 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
Number analyzed (Participants) | 34 | 32
Participants | 28 | 24

ADVERSE EVENTS:
Time Frame: From first dose up to 28 weeks
Description: Safety population included all participants who received at least one dose of study drug. Participants were summarized according to study drug regimen received.
Arm/Group | CTP-543 12 mg BID | CTP-543 24 mg QD
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/32
Other Adverse Events (participants affected / at risk) | 28/34 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTP-543 12 mg BID (N=34) | CTP-543 24 mg QD (N=32)
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTP-543 12 mg BID (N=34) | CTP-543 24 mg QD (N=32)
Palpitations (Cardiac disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 1
Seasonal allergy (General disorders) | 2 | 0
Folliculitis (General disorders) | 0 | 3
Nasopharyngitis (General disorders) | 4 | 3
Sinusitis (General disorders) | 2 | 0
Upper respiratory tract infection (General disorders) | 4 | 6
Urinary tract infection (General disorders) | 1 | 3
Alanine aminotransferase increased (Investigations) | 2 | 0
Amylase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bicarbonate decreased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 11 | 4
Blood potassium increased (Investigations) | 3 | 2
Lipase increased (Investigations) | 4 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Weight increased (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 4 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03941548/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03941548/SAP_003.pdf